CLINICAL TRIAL: NCT05532540
Title: Herpesvirus Immunology in Solid Organ Transplant Recipients - Liver Transplant Study
Acronym: HISTORY
Status: Active, not recruiting | Type: Observational
Sponsor: Susanne Dam Nielsen, MD, DMSc (Other)
Collaborators: Technical University of Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Susanne Dam Nielsen, MD, DMSc, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-22039226; 0073947 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Cytomegalovirus Infections; Varicella Zoster Virus Infection; Liver Transplant; Complications
Keywords: Cytomegalovirus; Herpesvirus 3, Human; Liver Transplantation; T-Lymphocytes; Inflammation; Immunodominant Epitopes; Major Histocompatibility Complex
MeSH Terms: conditions — Cytomegalovirus Infections; Varicella Zoster Virus Infection; Chickenpox; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected and separated into peripheral blood mononuclear cells (PBMC) and plasma, both of which are stored in a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant recipients: All adults enlisted for liver transplantation at Copenhagen University Hospital - Rigshospitalet (N = around 60 per year) will be invited to participate regardless of indication for liver transplantation. These participants are expected to undergo a liver transplantation and will continue in the study after the procedure.

SUMMARY:
Liver transplantation is the only curative treatment of end-stage liver disease, and every year, around 60 patients undergo liver transplantation in Denmark. Immunosuppressive therapy is necessary to avoid rejection of the transplanted organ.

Over 90% of adults have been infected with at least one herpesvirus, and it is characteristic for herpesviruses that after a first-time infection, the virus remains dormant in the body and may reactivate, particularly if the host is immunosuppressed. An effective immune response against reactivation depends highly on T cells, but T cells are suppressed by immunosuppressive drugs given to organ transplant recipients. Infections caused by herpesviruses are therefore very common in organ transplant recipients, and particularly two herpesviruses, cytomegalovirus (CMV) and varicella-zoster virus (VZV) pose challenges after transplantation.

CMV causes significant morbidity in transplant recipients, contributes to increased mortality and may contribute to loss of the transplanted organ. CMV infections occur in around 40% of liver transplant recipients within a year of transplantation. VZV causes chickenpox at first-time infection and shingles at reactivation. VZV is the second-most common infection in transplant recipients and occurs in around 9% of liver transplant recipients each year. Organ transplant recipients are at higher risk for disseminated disease with complications compared to immunocompetent persons.

A limited number of drugs exist that reduce the risk of and treat CMV infection, but they may cause significant adverse events, and drug resistance is emerging. To avoid CMV infection, some liver transplant recipients receive prophylactic therapy, but due to toxicity, new treatment modalities are warranted. This requires knowledge about herpesvirus specific T cell function in liver transplant recipients, which currently is limited.

The aim of this study is to provide an in-depth description of the protective immune response and immunological risk factors for CMV and VZV infections in liver transplant recipients and to identify patients at high risk in order to provide a platform for future treatment modalities against CMV and VZV infections in liver transplant recipients.

DETAILED DESCRIPTION:
The Herpesvirus Immunology in Solid Organ Transplant Recipients - Liver Transplant Study (HISTORY) is a prospective cohort study that aims to provide in-depth characterisation of the protective immune response and immunological risk factors for CMV and VZV infections in liver transplant recipients and to identify patients at high risk of infection based on clinical and immunological risk factors. All adult patients enlisted for liver transplantation at the Copenhagen University Hospital - Rigshospitalet will be invited to participate regardless of indication for transplantation.

At study entry, participants will fill out a questionnaire regarding health and medication use. Blood samples will be collected at study entry when enlisted for transplantation, at pre-defined intervals after transplantation, and if primary infection with or reactivation of CMV or VZV occurs during follow-up. Health data will be collected from hospital records and national registries.

Blood samples will be separated into peripheral blood mononuclear cells (PBMC) and plasma and stored in a biobank for analysis of PBMC phenotype and function, concentrations of inflammatory markers and mediators, CMV and VZV viral load and serology and other in-depth immunological analyses. Analyses will be performed at the Technical University of Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Enlisted for liver transplantation at Copenhagen University Hospital - Rigshospitalet
* Aged 18 years or older

Exclusion Criteria:

* Inability to understand the study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults enlisted for liver transplantation at Copenhagen University Hospital - Rigshospitalet (N = around 60 per year) will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency, phenotype and function of CMV- and VZV-specific T cells (descriptive) | 1.5 years
  Including: TCR clonotypes, cell surface markers and cytokine profile of T cell populations specific towards immunodominant CMV and VZV epitopes.

SECONDARY OUTCOMES:
Primary CMV infection | 10 years
VZV reactivation | 10 years
CMV reactivation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne D Nielsen, Professor, MD, DMSc, Principal Investigator — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Sine R Hadrup, Professor, MSc, PhD, Principal Investigator — Department of Health Technology, Technical University of Denmark; Moises Alberto Suarez Zdunek, MD, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Sebastian R Hamm, BSc, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Annemette Hald, RN, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Sunil K Saini, MSc, PhD, Study Director — Department of Health Technology, Technical University of Denmark; Allan Rasmussen, MD, Study Director — Department of Surgical Gastroenterology, Copenhagen University Hospital - Rigshospitalet; Jens G Hillingsø, MD, PhD, Study Director — Department of Surgical Gastroenterology, Copenhagen University Hospital - Rigshospitalet; Christian R Pedersen, MD, Study Director — Department of Surgical Gastroenterology, Copenhagen University Hospital - Rigshospitalet
Locations (3):
- Denmark (3):
  - Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Department of Surgical Gastroenterology, Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Department of Health Technology, Technical University of Denmark, Lyngby

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suarez-Zdunek MA, Saini SK, Pedersen CR, Hamm SR, Hald A, Rasmussen A, Hillingso JG, Hadrup SR, Nielsen SD. Herpesvirus immunology in solid organ transplant recipients - liver transplant study (HISTORY): a retrospective and prospective observational cohort study. BMC Infect Dis. 2023 Apr 6;23(1):214. doi: 10.1186/s12879-023-08153-8. PMID 37024811